CLINICAL TRIAL: NCT03970330
Title: A Randomized Double-Blind Placebo-Controlled Trial to Assess the Effectiveness of Low-Dose Naltrexone in Combination With Standard Treatment in Women With Chronic Pelvic Pain Secondary to Endometriosis
Brief Title: Low-Dose Naltrexone in Combination With Standard Treatment in Women With Endometriosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Original PI left institution, lack of funding to continue
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kristin Riley, MD, Asst. Professor of Obstetrics and Gynecology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Study00011187
Record Dates: First submitted 2019-05-15; First posted 2019-05-31 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Endometriosis
Keywords: endometriosis; pelvic pain; opioid; narcotic
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Naltrexone; Norethindrone Acetate

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low-Dose Naltrexone (Experimental): 12-week intervention period of 4.5 mg daily naltrexone in combination with standard treatment of 5-15 mg daily norethindrone acetate
  Interventions: Drug: Naltrexone; Drug: Norethindrone Acetate
- Placebo (Placebo Comparator): 12-week intervention period of daily placebo in combination with standard treatment of 5-15 mg daily norethindrone acetate
  Interventions: Drug: Norethindrone Acetate; Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 4.5mg daily dose, taken orally
  Other Names: REVIA
  Arms: Low-Dose Naltrexone
Drug: Norethindrone Acetate — 5 - 15mg daily dose, taken orally
Drug: Placebo — daily placebo pill, taken orally
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if the addition of Low Dose Naltrexone to standard endometriosis treatments will improve patient reported endometriosis associated pain.

DETAILED DESCRIPTION:
The central hypothesis of the research study is that low dose naltrexone (LDN), in combination with hormonal suppression of endometriosis (standard of care), will lead to significant improvement of endometriosis-related pain.

The proposal seeks to:

1. determine if the addition of LDN to standard endometriosis treatments will improve patient- reported endometriosis associated pain using daily Visual Analogue Scale (VAS) scores and
2. measure the impact of treatment on quality of life as measured by validated questionnaires including the Endometriosis Health Profile-30 (EHP30) and the Patient's Global Impression of Change (PGIC).

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female ages 18 to 45 years old on the day of signing informed consent.
* Must agree to use only study-specific analgesic medications during the study and is not known to be intolerant to them.
* Diagnosed with endometriosis and has had, within the last 10 years prior to signing the informed consent, surgical diagnosis with direct visualization and/or histopathologic confirmation of endometriosis.
* Is not expected to undergo gynecological surgery or other surgical procedures for treatment of endometriosis during the study period.
* Agrees to use contraception if not surgically sterile during the entire study.
* Patients using oral contraceptives, LARCs and/or GnRH agonists/antagonists for contraception and/or management of endometriosis, with a stable regimen, will be able to continue in the study, however, women using oral contraceptives and GnRH agonist/antagonists will be switched to Norethindrone acetate during the 1-2 week run-in period as prescribed by principle investigator.

Exclusion Criteria:

* Women that are pregnant, breastfeeding or trying to conceive.
* Patients with chronic daily narcotic use and any chronic pain or frequently reoccurring pain condition, other than endometriosis, that is treated with opioids or requires analgesics for more than 7 days per month.
* Patients with abnormal liver function tests (greater than 3x normal limit) in the past year or history of liver disease. Routine screening of liver function is not required.
* Non-English speaking or inability to read and understand English secondary, in part, to the need to read and report daily results in English.
* Undiagnosed vaginal bleeding
* Patients with history of opioid, illicit drug or alcohol abuse
* Patients currently taking thioridazine
* Patients with a history of suicidality
* Patients with current or history of unstable depression or other psychiatric disorder who, by PI judgement, are unstable or not well controlled
* Known, suspected or history of cancer of the breast
* Active deep vein thrombosis, pulmonary embolism or history of these conditions
* Active or recent arterial thromboembolic disease (e.g., stroke, myocardial infarction)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Endometriosis is specifically associated to females.
Enrollment: 9 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Riley, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared that underlie the results reported in this article, after deidentification. Documents that will be available are the study protocol, statistical analysis plan, informed consent. Analyses is to achieve the study aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available one year after publication according to PMCID journal guidelines.
Access Criteria: Data will plan to be published in a peer-reviewed journal and /or posted at clinicaltrials.gov websites or other websites per request of the NIH. Materials will also be accessible through email contact of Primary Investigator.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Dose Naltrexone | Placebo
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose Naltrexone | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (9) | 27.5 (3.4) | 28.9 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Score Area Under the Curve (AUC)
Description: Pain is reported daily using the Visual Analog Scale, a 100mm horizontal line on which the patient's pain intensity is represented by a point between the extremities of 0 (no pain) and 100 (worst pain). The final outcome measure will be calculated as area under the curve from randomization through 12-weeks of intervention. AUC was calculated using the trapezoid rule. Calculated AUC per subject across this 12-week period can range from 0 - 8300.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale*days
Arm/Group | Low-Dose Naltrexone | Placebo
Number analyzed (Participants) | 5 | 4
units on a scale*days | 2461 (1445) | 1338 (697)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone vs Placebo; Test type: Superiority; p = 0.20, t-test, 2 sided; Mean Difference (Final Values) = 1123, 95% CI 2-sided [-755 to 3000] — Difference calculated as Naltrexone minus Placebo

2. Secondary Outcome: EHP-30 Score
Description: Quality of life measured by the validated Endometriosis Health Profile (EHP-30) questionnaire. Scores range from 0 (best health status) to 100 (worst health status).
Time Frame: Baseline, 4, 8, 12, and 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-Dose Naltrexone | Placebo
Number analyzed (Participants) | 5 | 4
score on a scale
  Baseline | 56.5 (18.3) | 27.6 (19.4)
  Week 4 | 35.5 (16.6) | 25.1 (17.1)
  Week 8 | 34.9 (22.8) | 16.0 (8.0)
  Week 12 | 34.1 (26.6) | 18.6 (15.8)
  Week 16 | 35.7 (28.0) | 28.9 (23.3)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at BASELINE; Test type: Superiority; p = 0.06, Mixed Models Analysis; A single model was run with comparisons between naltrexone and placebo at each visit (not adjusted for multiple comparisons); Mean Difference (Final Values) = 28.9, 95% CI 2-sided [-1.9 to 59.6] — Difference calculated as Naltrexone minus Placebo
Statistical Analysis 2: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 4; Test type: Superiority; p = 0.48, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 10.4, 95% CI 2-sided [-20.3 to 41.2] — Difference calculated as Naltrexone minus Placebo
Statistical Analysis 3: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 8; Test type: Superiority; p = 0.21, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 18.9, 95% CI 2-sided [-11.8 to 49.6] — Difference calculated as Naltrexone minus Placebo
Statistical Analysis 4: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 12; Test type: Superiority; p = 0.30, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 15.5, 95% CI 2-sided [-15.2 to 46.2] — Difference calculated as Naltrexone minus Placebo
Statistical Analysis 5: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 16; Test type: Superiority; p = 0.65, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-24.0 to 37.5] — Difference calculated as Naltrexone minus Placebo

3. Secondary Outcome: PGIC Score (Painful Periods)
Description: Patient's Global Impression of Change (PGIC) scale will be used to rate painful periods. This is a 7 point scale ranging from 1 (much worse) to 7 (much better).
Time Frame: 4, 8, 12 and 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Low-Dose Naltrexone | Placebo
Number analyzed (Participants) | 5 | 4
units on a scale
  4 weeks | 4.0 [4.0 to 4.0] | 6.5 [5.5 to 7.0]
  8 weeks | 4.0 [4.0 to 4.0] | 6.5 [5.5 to 7.0]
  12 weeks | 4.0 [4.0 to 4.0] | 6.5 [6.0 to 7.0]
  16 weeks | 4.0 [4.0 to 5.0] | 4.5 [4.0 to 5.5]
Statistical Analysis 1: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 4; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 8; Test type: Superiority; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 12; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 16; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: PGIC Score (Nonmenstrual Pelvic Pain)
Description: Patient's Global Impression of Change (PGIC) scale will be used to rate nonmenstrual pelvic pain. This is a 7 point scale ranging from 1 (much worse) to 7 (much better).
Time Frame: 4, 8, 12 and 16 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Low-Dose Naltrexone | Placebo
Number analyzed (Participants) | 5 | 4
units on a scale
  Week 4 | 5.0 [4.0 to 6.0] | 6.5 [5.5 to 7.0]
  Week 8 | 4.0 [4.0 to 6.0] | 6.5 [5.5 to 7.0]
  Week 12 | 4.0 [4.0 to 6.0] | 6.5 [6.0 to 7.0]
  Week 16 | 4.0 [4.0 to 6.0] | 5.5 [4.5 to 6.0]
Statistical Analysis 1: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treament groups at WEEK 4; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 8; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 12; Test type: Superiority; p = 0.20, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 16; Test type: Superiority; p = 0.53, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: PGIC Score (Dyspareunia)
Description: Patient's Global Impression of Change (PGIC) scale will be used to rate pelvic pain during sex. This is a 7 point scale ranging from 1 (much worse) to 7 (much better).
Time Frame: 4, 8, 12 and 16 weeks
Population: This measure was only assessed in patients who had intercourse during study treatment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Low-Dose Naltrexone | Placebo
Number analyzed (Participants) | 2 | 3
units on a scale
  Week 4 | 4.0 [4.0 to 4.0] | 6.0 [4.0 to 6.0]
  Week 8 | 4.0 [4.0 to 4.0] | 6.0 [4.0 to 7.0]
  Week 12 | 4.0 [4.0 to 4.0] | 6.0 [4.0 to 6.0]
  Week 16 | 4.0 [4.0 to 4.0] | 5.0 [4.0 to 7.0]
Statistical Analysis 1: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 4; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 8; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 12; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Low-Dose Naltrexone vs Placebo; Comparison of treatment groups at WEEK 16; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Ibuprofen Use
Description: Average # of ibuprofen 200 mg pills per week during the study treatment period
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pills/week
Arm/Group | Low-Dose Naltrexone | Placebo
Number analyzed (Participants) | 5 | 4
pills/week | 5.5 (3.9) | 1.2 (1.3)
Statistical Analysis 1: Comparison: Low-Dose Naltrexone vs Placebo; Test type: Superiority; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [-0.6 to 9.2] — Difference calculated as Naltrexone minus Placebo

7. Secondary Outcome: Oxycodone Use
Description: Number of subjects who used oxycodone at any time during the study
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low-Dose Naltrexone | Placebo
Number analyzed (Participants) | 5 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse event collection occurred every 4 weeks (during study visits).
Arm/Group | Low-Dose Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 3/5 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Naltrexone (N=5) | Placebo (N=4)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Poison Ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin sensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Strep throat (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1)
Night sweats (General disorders) | 2 (2) | 1 (1)
Vivid dreams (General disorders) | 1 (1) | 0 (0)
Headaches (General disorders) | 1 (1) | 0 (0)
Leg contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03970330/Prot_SAP_000.pdf